CLINICAL TRIAL: NCT02454075
Title: A Pilot Trial of YF476, a Gastrin Antagonist, in Patients With Type II Gastric Carcinoids Associated With Zollinger-Ellison Syndrome
Brief Title: YF476 and Type II Gastric Carcinoids
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Trio Medicines Ltd. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-010; 11-DK-0114 (Other: NIHR); NCT01322542 (obsolete NCT alias)
Record Dates: First submitted 2015-05-13; First posted 2015-05-27 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Zollinger-Ellison Syndrome
Keywords: YF476; netazepide; gastric carcinoids; Zollinger-Ellison syndrome
MeSH Terms: conditions — Zollinger-Ellison Syndrome | interventions — YF 476

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eligible patients (Experimental): The dose will be 100 mg YF476 once daily. When 6 patients have completed 12 weeks' treatment with that dose, it may be increased to 150 or 200 mg once daily. Patients will have type II gastric carcinoids and/or ECL cell hyperplasia/dysplasia.
  Interventions: Drug: YF476

INTERVENTIONS:
Drug: YF476 — Gastrin receptor antagonist
  Other Names: Netazepide

SUMMARY:
This study will evaluate whether treatment with YF476 is safe and effective in reducing the size of type II gastric carcinoid tumours, or limiting the abnormal growth of gastric ECL cells, in patients with Zollinger-Ellison syndrome.

ELIGIBILITY:
Inclusion criteria:

1. Men; post-menopausal women; pre-menopausal women who have been sterilised by tubal ligation, hysterectomy or bilateral oophorectomy; or pre-menopausal women using one of the allowed methods of contraception: condom and spermicide or intra-uterine device.
2. Patients with serum gastrin >250 pg/mL.
3. Hepatic function: AST and ALT ≤2.0 x ULN; total bilirubin ≤1.0 x ULN.
4. Renal function: serum creatinine <1.0 x ULN.
5. Haematologic function: Hb ≥10.0 g/dL; WBC ≥3.5 x 10e9 /L; ANC ≥1.5 x 10e9 /L; platelets ≥100 x 10e9 /L.
6. Coagulation parameters: INR or PT ≤1.0 x ULN; PTT ≤1.0 x ULN.
7. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
8. Willingness to give fully-informed, written consent.

Exclusion criteria:

1. Patients under 18 years.
2. Women who are pregnant, lactating or using a steroid contraceptive.
3. Prior gastric resection or bypass.
4. Planned gastrinoma resection during the study period.
5. Patients on somatostatin analogues, except for those on therapy for >6 months with stable or worsening carcinoids.
6. Inability to tolerate endoscopy, or refusal of endoscopy.
7. Physical findings, ECG (especially prolonged QTc interval >450 msec), or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the subject.
8. Certain medicines and herbal remedies taken during the 7 days before visit 2.
9. Participation in a trial of an IMP within the previous 28 days.
10. Presence of drug or alcohol abuse.
11. History or baseline findings of:

    * type 1 diabetes mellitus;
    * pancreatitis (baseline amylase and/or >2.0 x ULN);
    * hepatitis B, hepatitis C or HIV;
    * malabsorption syndrome or inability to swallow or retain oral medicine;
    * major surgery <28 days prior to enrolment;
    * ECOG performance status >2; or
    * another cancer within 3 years except for basal carcinoma of the skin or cervical carcinoma in-situ.
    * Also, any clinically significant and uncontrolled major morbidity including but not limited to; serious cardiac disease (unstable angina, s/p myocardial infarction <1 month); respiratory disease (advanced COPD or pulmonary fibrosis); uncontrolled hypertension; or active systemic infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-04-11 (Actual); Primary Completion 2012-06-22 (Actual); Study Completion 2012-06-22 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Eligible Patients: Patients received 100 mg YF476 orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Eligible Patients
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eligible Patients
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
Serum gastrin [Number; unit: pg/mL] — Measured on screening visit
  pg/mL
    Patient 01 | 587
    Patient 02 | 11348
    Patient 03 | 1393
Serum chromagraninA (CgA) [Number; unit: ng/mL] — Measured pre-dose on Day 1, Visit 2
  ng/mL
    Patient 01 | 3410
    Patient 02 | 11200
    Patient 03 | 2430
Size of gastric carcinoids [Mean (Full Range); unit: mm^2] — Measured via endoscopy on Visit 2
  mm^2
    Patient 01 | 54.79 [29.68 to 74.92]
    Patient 02 | 70.20 [37.09 to 131.21]
    Patient 03 | 24.77 [12.00 to 34.95]

OUTCOME MEASURES:

1. Primary Outcome: Regression of Gastric Carcinoids and/or ECL Cell Hyperplasia Defined by Physical Measurements Taken During Endoscopy
Description: Regression is defined as a 25% reduction in the size / number of endoscopically evident type II gastric carcinoids. For each participant, three gastric carcinoids were identified and measured at baseline. The same gastric carcinoids were then measured at the Week 12 visit and the percentage difference in size from baseline calculated. The mean percentage change of the three gastric carcinoids per participant is recorded.
Time Frame: Week 12 visit
Population: The mean percentage decrease in three gastric carcinoids (measured at Week 12 visit) compared with baseline.
Measure: Mean (Standard Deviation); unit: percentage decrease in carcinoid size
Arm/Group | Eligible Patients
Number analyzed (Participants) | 3
percentage decrease in carcinoid size
  Patient 01, Week 12 visit: number analyzed (Participants) | 1
  Patient 01, Week 12 visit | 23.7 (6.23)
  Patient 02, Week 12 visit: number analyzed (Participants) | 1
  Patient 02, Week 12 visit | 8.6 (26.96)
  Patient 03, Week 12 visit: number analyzed (Participants) | 1
  Patient 03, Week 12 visit | 10.8 (24.44)

2. Primary Outcome: A Reduction of 25% in the Gastric ECL Cell Density.
Description: A reduction of 25% in the gastric ECL cell density.
Time Frame: Week 12 visit
Population: Due to the early termination of the study, the data for this outcome measure were not collected.
Arm/Group | Eligible Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Improvement in Histological Grade of Gastric Carcinoids/ECL Cell Hyperplasia Defined by Physical Measurements Taken During Endoscopy
Description: Reduction in the histological grade of the carcinoids/hyperplasia when compared to baseline.
Time Frame: Week 12 visit
Population: Due to the early termination of the study, the data for this outcome measure were not collected.
Arm/Group | Eligible Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Level of Chromogranin A (CgA) Biomarkers Measured in Blood Samples
Description: The level of a key biomarker chromogranin A (CgA) that is circulating in the blood was measured.
Time Frame: Week 6 visit, Week 12 visit, Follow-up (12 weeks after stopping YF476 treatment)
Population: The CgA data is provided for each participant at each visit
Measure: Number; unit: ng/mL
Arm/Group | Eligible Patients
Number analyzed (Participants) | 3
ng/mL
  Patient 01, Week 6 visit: number analyzed (Participants) | 1
  Patient 01, Week 6 visit | 2600
  Patient 01, Week 12 visit: number analyzed (Participants) | 1
  Patient 01, Week 12 visit | 2700
  Patient 01, Follow-up: number analyzed (Participants) | 1
  Patient 01, Follow-up | 12300
  Patient 02, Week 6 visit: number analyzed (Participants) | 1
  Patient 02, Week 6 visit | 11950
  Patient 02, Week 12 visit: number analyzed (Participants) | 1
  Patient 02, Week 12 visit | 15350
  Patient 02, Follow up: number analyzed (Participants) | 1
  Patient 02, Follow up | 24100
  Patient 03, Week 6 visit: number analyzed (Participants) | 1
  Patient 03, Week 6 visit | 213
  Patient 03, Week 12 visit: number analyzed (Participants) | 1
  Patient 03, Week 12 visit | NA — Sample taken but source documentation not provided
  Patient 03, Follow-up: number analyzed (Participants) | 1
  Patient 03, Follow-up | NA — Sample taken but source documentation not provided

5. Secondary Outcome: Acid Control Study 1, Control of Gastric Acid Secretion Assessed by Changes in Drug-controlled Gastric Acid Analysis, Volume of Gastric Aspirate
Description: Assessed by changes in drug-controlled gastric acid analysis. A nasogastric tube (NGT) was placed through one nare and into the stomach. Gastric secretions were suctioned and discarded at T = 0 and then aspirated for 1 h in 15 min increments to measure the control acid output. Patients who could not tolerate NGT placement had endoscopic gastric analysis (EGA) performed during upper endoscopy. During EGA, a single 10 - 15 min collection was aspirated under direct visualization. Patients 01 and 02 had acid measured via NGT, whereas Patient 03 had acid measured via EGA. At the Week 2 visit, the baseline acid control was measured. At the Week 6 visit, the acid control was measured after a dose of netazepide. Results are provided for three acid control measures:
  1. Volume of aspirate (mL)
  2. Acid in aspirate (mEq)
  3. Acid output (mEq)
Time Frame: Week 2 visit (baseline) and Week 6 visit
Population: Patients had the volume of gastric aspirate measured at Week 2 and Week 6 visit, by either nasogastric tube (NGT; Patient 01 and Patient 02) or endoscopic gastric analysis (EGA; Patient 03). Data is provided for each visit and participant.
Measure: Number; unit: mL
Groups:
- Eligible Patients: The dose will be an oral dose of 100 mg YF476 once daily for 12 weeks. When 6 patients have completed 12 weeks' treatment with that dose, it may be increased to 150 or 200 mg once daily. Patients will have type II gastric carcinoids and/or ECL cell hyperplasia/dysplasia.
  YF476: Gastrin receptor antagonist
Arm/Group | Eligible Patients
Number analyzed (Participants) | 3
mL
  Patient 01, Week 2 visit, Day 1, 0 - 15 min: number analyzed (Participants) | 1
  Patient 01, Week 2 visit, Day 1, 0 - 15 min | 12
  Patient 01, Week 2 visit, Day 1, 15 - 30 min: number analyzed (Participants) | 1
  Patient 01, Week 2 visit, Day 1, 15 - 30 min | 10
  Patient 01, Week 2 visit, Day 1, 30 - 45 min: number analyzed (Participants) | 1
  Patient 01, Week 2 visit, Day 1, 30 - 45 min | 4
  Patient 01, Week 2 visit, Day 1, 45 - 60 min: number analyzed (Participants) | 1
  Patient 01, Week 2 visit, Day 1, 45 - 60 min | 15
  Patient 01, Week 6 visit, Day 1, 0 - 15 min: number analyzed (Participants) | 1
  Patient 01, Week 6 visit, Day 1, 0 - 15 min | 5
  Patient 01, Week 6 visit, Day 1, 15 - 30 min: number analyzed (Participants) | 1
  Patient 01, Week 6 visit, Day 1, 15 - 30 min | 7
  Patient 01, Week 6 visit, Day 1, 30 - 45 min: number analyzed (Participants) | 1
  Patient 01, Week 6 visit, Day 1, 30 - 45 min | 17
  Patient 01, Week 6 visit, Day 1, 45 - 60 min: number analyzed (Participants) | 1
  Patient 01, Week 6 visit, Day 1, 45 - 60 min | 7
  Patient 02, Week 2 visit, Day 1, 0 - 15 min: number analyzed (Participants) | 1
  Patient 02, Week 2 visit, Day 1, 0 - 15 min | 10
  Patient 02, Week 2 visit, Day 1, 15 - 30 min: number analyzed (Participants) | 1
  Patient 02, Week 2 visit, Day 1, 15 - 30 min | 5
  Patient 02, Week 2 visit, Day 1, 30 - 45 min: number analyzed (Participants) | 1
  Patient 02, Week 2 visit, Day 1, 30 - 45 min | 40
  Patient 02, Week 2 visit, Day 1, 45 - 60 min: number analyzed (Participants) | 1
  Patient 02, Week 2 visit, Day 1, 45 - 60 min | 25
  Patient 02, Week 6 visit, Day 1, 0 - 15 min: number analyzed (Participants) | 1
  Patient 02, Week 6 visit, Day 1, 0 - 15 min | 30
  Patient 02, Week 6 visit, Day 1, 15 - 30 min: number analyzed (Participants) | 1
  Patient 02, Week 6 visit, Day 1, 15 - 30 min | 50
  Patient 02, Week 6 visit, Day 1, 30 - 45 min: number analyzed (Participants) | 1
  Patient 02, Week 6 visit, Day 1, 30 - 45 min | 10
  Patient 02, Week 6 visit, Day 1, 45 - 60 min: number analyzed (Participants) | 1
  Patient 02, Week 6 visit, Day 1, 45 - 60 min | 10
  Patient 02, Week 6 visit, Day 1, 60 - 75 min: number analyzed (Participants) | 1
  Patient 02, Week 6 visit, Day 1, 60 - 75 min | 49
  Patient 03, Week 2 visit, Day 1, 0 - 15 min: number analyzed (Participants) | 1
  Patient 03, Week 2 visit, Day 1, 0 - 15 min | 15
  Patient 03, Week 6 visit, Day 1, 0 - 15 min: number analyzed (Participants) | 1
  Patient 03, Week 6 visit, Day 1, 0 - 15 min | 17

6. Secondary Outcome: Decrease in ECL Cell-specific Products Assessed by Quantitative PCR
Description: Assessed by quantitative PCR.
Time Frame: Week 2 visit (baseline), Week 6 visit, Week 12 visit, Follow-up (12 weeks after stopping YF476 treatment)
Population: Data was not collect due to early termination of the study.
Arm/Group | Eligible Patients
Number analyzed (Participants) | 0

7. Secondary Outcome: Improvement in Reflux/Dyspepsia Symptoms Using the Gastroesophageal Reflux Disease Health Related Quality of Life (GERD-HRQL) Instrument
Description: Assessed by the Gastroesophageal Reflux Disease Health Related Quality of Life (GERD-HRQL) instrument. Patients assessed a total of 10 symptoms on a scale of 0-5 where: 0 = no symptoms; 1 = symptoms noticeable, but not bothersome; 2 = symptoms noticeable and bothersome, but not every day; 3 = symptoms bothersome everyday; 4 = symptoms affect daily activities; and 5 = symptoms are incapacitating (unable to do daily activities). The total score was summed and reported. The maximum obtainable total score was 50 and minimum obtainable total score was 0, with higher scores indicating a worse outcome and lower scores indicating a better outcome.
Time Frame: Week 2 visit (baseline), Week 6 visit, Week 12 visit, Follow-up (12 weeks after stopping YF476 treatment)
Population: For each patient, the total score on the GERD-HRQL assessment questionnaire at each visit was summed and reported. Data is provided for each visit and participant.
Measure: Number; unit: score on a scale
Arm/Group | Eligible Patients
Number analyzed (Participants) | 3
score on a scale
  Patient 1, Week 2 visit: number analyzed (Participants) | 1
  Patient 1, Week 2 visit | 3
  Patient 1, Week 6 visit: number analyzed (Participants) | 1
  Patient 1, Week 6 visit | 3
  Patient 1, Week 12 visit: number analyzed (Participants) | 1
  Patient 1, Week 12 visit | 2
  Patient 1, Follow up visit: number analyzed (Participants) | 1
  Patient 1, Follow up visit | 4
  Patient 2, Week 2 visit: number analyzed (Participants) | 1
  Patient 2, Week 2 visit | 0
  Patient 2, Week 6 visit: number analyzed (Participants) | 1
  Patient 2, Week 6 visit | 26
  Patient 2, Week 12 visit: number analyzed (Participants) | 1
  Patient 2, Week 12 visit | 10
  Patient 2, Follow up visit: number analyzed (Participants) | 1
  Patient 2, Follow up visit | 19
  Patient 3, Week 2 visit: number analyzed (Participants) | 1
  Patient 3, Week 2 visit | 0
  Patient 3, Week 6 visit: number analyzed (Participants) | 1
  Patient 3, Week 6 visit | 0
  Patient 3, Week 12 visit: number analyzed (Participants) | 1
  Patient 3, Week 12 visit | 0
  Patient 3, Follow up visit: number analyzed (Participants) | 1
  Patient 3, Follow up visit | 0

8. Secondary Outcome: Safety and Tolerability
Description: Assessed by monitoring adverse events reported by patients
Time Frame: Week 2 visit (baseline), Week 6 visit, Week 12 visit, Follow-up (12 weeks after stopping YF476 treatment)
Measure: Number; unit: adverse events
Arm/Group | Eligible Patients
Number analyzed (Participants) | 3
adverse events
  Week 2 visit: number of treatment related adverse events | 0
  Week 6 visit: number of treatment related adverse events | 0
  Week 12 visit: number of treatment related adverse events | 0
  Follow up visit: number of treatment related adverse events | 0

9. Secondary Outcome: Circulating Plasma Concentration of Gastrin
Description: The level of gastrin biomarkers circulating in the blood was measured.
Time Frame: Week 6 visit, Week 12 visit, Follow-up (12 weeks after stopping YF476 treatment)
Population: Data is provided for each visit of each patient. Follow up data is missing for Patient 03 (samples were taken but results not provided).
Measure: Number; unit: pg/mL
Arm/Group | Eligible Patients
Number analyzed (Participants) | 3
pg/mL
  Patient 01, Week 6 visit: number analyzed (Participants) | 1
  Patient 01, Week 6 visit | 509
  Patient 01, Week 12 visit: number analyzed (Participants) | 1
  Patient 01, Week 12 visit | 355
  Patient 01, Follow-up: number analyzed (Participants) | 1
  Patient 01, Follow-up | 1105
  Patient 02, Week 6 visit: number analyzed (Participants) | 1
  Patient 02, Week 6 visit | 13049
  Patient 02, Week 12 visit: number analyzed (Participants) | 1
  Patient 02, Week 12 visit | 12846
  Patient 02, Follow-up: number analyzed (Participants) | 1
  Patient 02, Follow-up | 14113
  Patient 03, Week 6: number analyzed (Participants) | 1
  Patient 03, Week 6 | 706
  Patient 03, Week 12: number analyzed (Participants) | 1
  Patient 03, Week 12 | 718

10. Secondary Outcome: Acid Control Study 2, Control of Gastric Acid Secretion Assess by Changes in Drug-controlled Gastric Acid Analysis: Acid Content in Gastric Aspirate
Description: as for outcome 5
Time Frame: Week 2 visit (baseline) and Week 6 visit
Population: Patients had the acid content in gastric aspirate measured at Week 2 and Week 6 visit, by either nasogastric tube (NGT; Patient 01 and Patient 02) or endoscopic gastric analysis (EGA; Patient 03). Data is provided for each visit and participant.
Measure: Number; unit: mEq
Arm/Group | Eligible Patients
Number analyzed (Participants) | 3
mEq
  Patient 01, Week 2 visit, Day 1, 0 - 15 min: number analyzed (Participants) | 1
  Patient 01, Week 2 visit, Day 1, 0 - 15 min | 5.6
  Patient 01, Week 2 visit, Day 1, 15 - 30 min: number analyzed (Participants) | 1
  Patient 01, Week 2 visit, Day 1, 15 - 30 min | 4.9
  Patient 01, Week 2 visit, Day 1, 30 - 45 min: number analyzed (Participants) | 1
  Patient 01, Week 2 visit, Day 1, 30 - 45 min | 5.1
  Patient 01, Week 2 visit, Day 1, 45 - 60 min: number analyzed (Participants) | 1
  Patient 01, Week 2 visit, Day 1, 45 - 60 min | 4.9
  Patient 01, Week 6 visit, Day 1, 0 - 15 min: number analyzed (Participants) | 1
  Patient 01, Week 6 visit, Day 1, 0 - 15 min | 6.9
  Patient 01, Week 6 visit, Day 1, 15 - 30 min: number analyzed (Participants) | 1
  Patient 01, Week 6 visit, Day 1, 15 - 30 min | 6.5
  Patient 01, Week 6 visit, Day 1, 30 - 45 min: number analyzed (Participants) | 1
  Patient 01, Week 6 visit, Day 1, 30 - 45 min | 6.6
  Patient 01, Week 6 visit, Day 1, 45 - 60 min: number analyzed (Participants) | 1
  Patient 01, Week 6 visit, Day 1, 45 - 60 min | 6.7
  Patient 02, Week 2 visit, Day 1, 0 - 15 min: number analyzed (Participants) | 1
  Patient 02, Week 2 visit, Day 1, 0 - 15 min | 6.7
  Patient 02, Week 2 visit, Day 1, 15 - 30 min: number analyzed (Participants) | 1
  Patient 02, Week 2 visit, Day 1, 15 - 30 min | 7.4
  Patient 02, Week 2 visit, Day 1, 30 - 45 min: number analyzed (Participants) | 1
  Patient 02, Week 2 visit, Day 1, 30 - 45 min | 7.0
  Patient 02, Week 2 visit, Day 1, 45 - 60 min: number analyzed (Participants) | 1
  Patient 02, Week 2 visit, Day 1, 45 - 60 min | 7.6
  Patient 02, Week 6 visit, Day 1, 0 - 15 min: number analyzed (Participants) | 1
  Patient 02, Week 6 visit, Day 1, 0 - 15 min | 1.2
  Patient 02, Week 6 visit, Day 1, 15 - 30 min: number analyzed (Participants) | 1
  Patient 02, Week 6 visit, Day 1, 15 - 30 min | 1.2
  Patient 02, Week 6 visit, Day 1, 30 - 45 min: number analyzed (Participants) | 1
  Patient 02, Week 6 visit, Day 1, 30 - 45 min | 1.2
  Patient 02, Week 6 visit, Day 1, 45 - 60 min: number analyzed (Participants) | 1
  Patient 02, Week 6 visit, Day 1, 45 - 60 min | 1.2
  Patient 02, Week 6 visit, Day 1, 60 - 75 min: number analyzed (Participants) | 1
  Patient 02, Week 6 visit, Day 1, 60 - 75 min | 1.2
  Patient 03, Week 2 visit, Day 1, 0 - 15 min: number analyzed (Participants) | 1
  Patient 03, Week 2 visit, Day 1, 0 - 15 min | 4.9
  Patient 03, Week 6 visit, Day 1, 0 - 15 min: number analyzed (Participants) | 1
  Patient 03, Week 6 visit, Day 1, 0 - 15 min | 1.1

11. Secondary Outcome: Acid Control Study 3, Control of Gastric Acid Secretion Assess by Changes in Drug-controlled Gastric Acid Analysis: Acid Output
Description: as for outcome 5
Time Frame: Week 2 visit (baseline) and Week 6 visit
Population: Patients had acid output measured at Week 2 and Week 6 visit, by either nasogastric tube (NGT; Patient 01 and Patient 02) or endoscopic gastric analysis (EGA; Patient 03). Data is provided for each visit and participant.
Measure: Number; unit: mEq
Arm/Group | Eligible Patients
Number analyzed (Participants) | 3
mEq
  Patient 01, Week 2 visit, Day 1, 0 - 15 min | 0.1
  Patient 01, Week 2 visit, Day 1, 15 - 30 min | 0
  Patient 01, Week 2 visit, Day 1, 30 - 45 min | 0
  Patient 01, Week 2 visit, Day 1, 45 - 60 min | 0.2
  Patient 01, Week 6 visit, Day 1, 0 - 15 min | 0
  Patient 01, Week 6 visit, Day 1, 15 - 30 min | 0
  Patient 01, Week 6 visit, Day 1, 30 - 45 min | 0
  Patient 01, Week 6 visit, Day 1, 45 - 60 min | 0
  Patient 02, Week 2 visit, Day 1, 0 - 15 min | 0.2
  Patient 02, Week 2 visit, Day 1, 15 - 30 min | 0
  Patient 02, Week 2 visit, Day 1, 30 - 45 min | 0.7
  Patient 02, Week 2 visit, Day 1, 45 - 60 min | 0.4
  Patient 02, Week 6 visit, Day 1, 0 - 15 min | 1.8
  Patient 02, Week 6 visit, Day 1, 15 - 30 min | 4.1
  Patient 02, Week 6 visit, Day 1, 30 - 45 min | 1.2
  Patient 02, Week 6 visit, Day 1, 45 - 60 min | 0.7
  Patient 02, Week 6 visit, Day 1, 60 - 75 min | 1.6
  Patient 03, Week 2 visit, Day 1, 0 - 15 min | 1.2
  Patient 03, Week 6 visit, Day 1, 0 - 15 min | 4.6

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with that treatment.
Groups:
- Eligible Patients: The dose will be an oral dose of 100 mg YF476 once daily. for 12 weeks. When 6 patients have completed 12 weeks' treatment with that dose, it may be increased to 150 or 200 mg once daily. Patients will have type II gastric carcinoids and/or ECL cell hyperplasia/dysplasia.
  YF476: Gastrin receptor antagonist
Arm/Group | Eligible Patients
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eligible Patients (N=3)
Toothache (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Hypertension (Vascular disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Upper respiratory tract infections (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No